CLINICAL TRIAL: NCT06309498
Title: Residual Adrenal Function in Addison's Disease
Acronym: ADD-RES
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 05C307
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: blood test — 11 DOC levels will be measured in enrolled patients
  Other Names: 11 DOC measurement

SUMMARY:
The main aim of this study is to assess the role of 11-deoxycortisol as surrogate marker of Residual adrenal function.

11-deoxycortisol levels will be assessed in all recruited patients

DETAILED DESCRIPTION:
Addison's disease is an autoimmune disease characterized by inadequate secretion of cortisol and aldosteron by adrenal cortex as a consequence of progressive destruction of the adrenal gland. The absence of specific signs and symptoms could delay the diagnosis and treatment. Considering the importance of these two hormones, a not adequate treatment can result in Addisonian crisis and even be a cause of increased mortality.

Actually, diagnosis is based either on low basal cortisol levels or cortisol levels after Synacthen test (250 mcg) < 500 nmol/L.

Adrenal insufficiency (AI) is most of the time the inevitable end result of the autoimmune process, but some cases of partial recovery of adrenal function in a patient with autoimmune Addison's disease have been described.

Recent evidence shows that 5-30% of Addison's patients, also after many years of disease, maintain a residual endogenous corticosteroid production thanks to a partial adrenal cortex functionality, known as residual adrenal function (RAF).

Indeed, some studies show how the 3-15% of patients have detectable cortisol at Synacthen 250 mcg test, demonstrating that in one third of patients with long-standing disease, some RAF was still present.

The clinical significance of this RAF is unknown but potentially can reduce the need of hormone replacement, affecting the patient's quality of life. An approach to determine residual endogenous cortisol production may be the measurement of its precursor, 11-deoxycortisol (11DOC).

The main aim of this study is to assess the role of 11DOC as surrogate marker of RAF.

It is expected that 15% of our population have a RAF. In patients with RAF we expect significantly higher 11DOC values and at the same time a lower prevalence of Addisonian crisis with a higher prevalence of complications as diabetes mellitus, arterial hypertension, osteoporosis and infections caused by the overtreatment.

Meanwhile, in patients without RAF a higher rate of Addisonian crisis despite a higher dose of treatment is expected.

The possibility to map the RAF in patients on hydrocortisone substitutive therapy by the use of a single marker (11DOC) could be useful as it permits to have a more patient- based medical approach without having to carry out time consuming tests (e.g.Synacthen Test).

Despite the pharmacological approach actually Addison's patients have an impaired quality of life. For the AI treatment in adults, the Endocrine European Society's recommended daily glucocorticoid replacement dose (DGRD) is 15 to 25 mg hydrocortisone. Under-replacement may result in weight loss, hypotension, hyponatremia, and death. In contrast, glucocorticoids excess may cause metabolic complications and immune suppression.

If this hypothesis were confirmed it could be helpful to reduce the DGRD in patients with RAF, in order to minimize the incidence of complication of long-term therapy. On the other side, in patients without RAF, it could be useful to take more attention to reduce the risk of Addisonian's crisis.

Last but not least, finding a marker of RAF, as 11DOC, without having to perform further tests, could allow to reduce timing and costs for the single Addison's patient evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Autoimmune Addison's disease
* Informed consent

Exclusion Criteria:

- Drugs affecting immune system or steroids other than hydrocortisone or cortisone acetate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adul patients affected with Autoimmune Addison's Disease
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of RAF | baseline
  residual adrenal function

SECONDARY OUTCOMES:
prevalence of adrenal crisis | 24 months
  prevalence of adrenal crisis in relation to RAF

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Morelli, PHD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearce SHS, Gan EH, Napier C. MANAGEMENT OF ENDOCRINE DISEASE: Residual adrenal function in Addison's disease. Eur J Endocrinol. 2021 Feb;184(2):R61-R67. doi: 10.1530/EJE-20-0894. PMID 33306039
- [Background] Vulto A, Bergthorsdottir R, van Faassen M, Kema IP, Johannsson G, van Beek AP. Residual endogenous corticosteroid production in patients with adrenal insufficiency. Clin Endocrinol (Oxf). 2019 Sep;91(3):383-390. doi: 10.1111/cen.14006. Epub 2019 Jun 20. PMID 31059146